CLINICAL TRIAL: NCT03930667
Title: Hem-o-lok Clips Versus ıntracorporeal Knotting for Closure of the Appendix Stump in Laparoscopic Appendectomy: Prospective Randomized Study
Brief Title: Closure of the Appendix Stump in Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orhan Üreyen (Other)
Responsible Party: Sponsor-Investigator, Orhan Üreyen, Clinical expert in General Surgery,Principal Investigator, Bozyaka Training and Research Hospital
Organization: Bozyaka Training and Research Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 24.03.2015-no:3
Record Dates: First submitted 2019-04-21; First posted 2019-04-29 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Appendicitis, Surgery
Keywords: Appendicitis; Laparoscopic Surgery; Cost Effectiveness
MeSH Terms: conditions — Appendicitis | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clips (Active Comparator): Closure of the appendix stump with hem-o-lok clips
  Interventions: Procedure: clips
- knotting (Experimental): Closure of the appendix stump with intracorporal knotting.
  Interventions: Procedure: knotting

INTERVENTIONS:
Procedure: clips
  Arms: clips
Procedure: knotting
  Arms: knotting

SUMMARY:
Aimed to the study evaluate the superiority of intracorporal sutures and Hem-o-lok clips in terms of efficiency.

DETAILED DESCRIPTION:
Performed laparoscopic surgery for acute appendicitis. Appendiceal stump was closed by Hem-o-lok clips (Group I) and intracorporal knotting (Group II) in a randomize manner. Groups were compared for cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute appendicitis

Exclusion Criteria:

* under 18 years of age
* other patology in addition to appendiceal pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
cost effectiveness | 4 years
  cost of treatment from surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Orhan Ureyen, Principal Investigator — Health Sciences University, İzmir Bozyaka Training and Research Hospital, General Surgery Department, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2015-2019